CLINICAL TRIAL: NCT02465996
Title: Gastric Barrier Dysfunction of Functional Dyspepsia and Therapeutic Response to Puyuanhewei Detected by Endomicroscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015SDU-QILU-G02
Record Dates: First submitted 2015-06-01; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Dyspepsia
Keywords: barrier dysfunction; functional dyspepsia; Confocal Laser Endomicroscopic; therapeutic response
MeSH Terms: conditions — Dyspepsia | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- postprandial distress syndrome (PDS) (Other): FD patients fulfilled Rome III criteria were subclassified into postprandial distress syndrome (PDS) or epigastric pain syndrome (EPS).
  pCLE examination was performed in PDS patients, and then those who were willing to receive Puyuanhewei to treat FD were given 4 pills three times a day for 4 weeks after pCLE examination.
  Interventions: Device: pCLE examination; Drug: Puyuanhewei
- epigastric pain syndrome (EPS) (Other): pCLE examination was performed in EPS patients, and then those who were willing to receive Puyuanhewei to treat FD were given 4 pills three times a day for 4 weeks after pCLE examination.
  Interventions: Device: pCLE examination; Drug: Puyuanhewei

INTERVENTIONS:
Device: pCLE examination — All FD patients received pCLE examination.
  Other Names: prob-based confocal laser endomicroscopy examination
Drug: Puyuanhewei — FD patients willing to receive Puyuanhewei were given 4 pills three times a day regardless of PDS or EPS for 4 weeks after pCLE examination.
  Other Names: Puyanhewei capsule administration

SUMMARY:
Functional dyspepsia might have impaired gastric mucosal dysfunction and Puyuanhewei may be helpful to improve the symptoms of FD.

DETAILED DESCRIPTION:
This study aimed to investigate the gastric mucosal dysfunction in functional dyspepsia (FD) and verify the efficacy of Puyuanhewei for treating FD and assess the relationship between gastric microalterations and therapeutic response by endomicroscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive outpatients aged 18 to 75 years old.
2. FD patients defined by the Rome III classification.
3. Willing to choose pCLE and no organic diseases.

Exclusion Criteria:

1. Severe liver, heart, or kidney diseases.
2. Current or past evidence of uncontrolled diabetes mellitus, psychosomatic disorders, such as depressive and anxiety disorders, and drug or alcohol abuse.
3. Pregnant or breastfeeding women.
4. Inability to give informed consent.
5. Use of nonsteroidal anti-inflammatory drugs, proton pump inhibitors, H2-receptor antagonists, antacids, prokinetics, or other injurious drugs (antibiotics, and steroids) in the prior two weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
pCLE score | within 1 hour after pCLE examination
  Used to assess the gastric barrier dysfunction of FD patients

SECONDARY OUTCOMES:
Leeds dyspepsia questionaire | baseline and 4th week
  Used to describe the change of severity of FD from baseline to the 4th week during the treatment
Main dyspepsia symptom score | baseline and 4th weeks
  Used to describe the change of severity and frequency of despepsia symptoms from baseline to the 4th week during the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China